CLINICAL TRIAL: NCT06761131
Title: Comparative Study Between Incidence of Linezolid-Induced Thrombocytopenia in Patients With Normal Renal Function Versus Patients With Impaired Renal Function
Brief Title: Compare Linezolid-Induced Thrombocytopenia in Patients With Normal Renal Function Versus Impaired Renal Function
Acronym: LinezRenal
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD35/2024
Record Dates: First submitted 2024-12-26; First posted 2025-01-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Thrombocytopaenia; Impaired Renal Function
MeSH Terms: conditions — Thrombocytopenia; Renal Insufficiency | interventions — Linezolid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group N (will be with normal renal function)
  Interventions: Drug: Linezolid (LZD)
- Group I (will be with impaired renal function)
  Interventions: Drug: Linezolid (LZD)

INTERVENTIONS:
Drug: Linezolid (LZD) — compare the incidence and magnitude of Linezolid induced thrombocytopenia

SUMMARY:
Linezolid exhibits a broad spectrum of activity against Gram-positive bacteria, including methicillin-resistant staphylococcus aureus (MRSA) and vancomycin-resistant enterococci. The major adverse effect associated with linezolid treatment is reversible myelosuppression, mostly thrombocytopenia. Recent studies have reported that the incidence of linezolid-induced thrombocytopenia was higher among patients with renal failure than in patients with normal renal function, although the underlying mechanisms explaining this toxicity are still unknown.

DETAILED DESCRIPTION:
Linezolid is an oxazolidinone antibiotic with the availability of intravenous and oral formulations. The latter has nearly 100% bioavailability and is expected to facilitate the treatment of infections caused by these organisms (Gram-positive bacteria).

In addition, linezolid has very favorable rates of penetration into tissues. This suggests a potential pharmacokinetic advantage of linezolid over glycopeptides in the treatment of deep-seated infections such as pneumonia and CNS infections.

Prolonged use of linezolid can lead to hematological side effects, particularly thrombocytopenia. Indeed, several studies have reported that the incidence of thrombocytopenia associated with linezolid therapy is much higher (7.5%-64.7%) than the incidence reported in an early clinical study (2.4%) conducted by the manufacturer.

Thrombocytopenia is a common complication in the intensive care unit (ICU), and its incidence ranges from 13 to 60 %.

Thrombocytopenia is defined as a platelet count of less than 100,000/μl or a decrease of at least 50 % from baseline. Thrombocytopenia can be characterized as mild (≥ 50,000/μl), moderate (30,000/μl to 50,000/μl) and severe (< 30,000/μl).

There are different causes of thrombocytopenia in critically ill patients: sepsis, severe malnutrition, neoplastic infiltration of bone marrow, radiation therapy, mechanical intravascular devices, autoimmune disorders, and the administration of heparin (heparin-induced thrombocytopenia, HIT).

Moreover, many drugs can cause thrombocytopenia. The incidence of drug-induced thrombocytopenia (DIT) is not well defined but is estimated to be at least ten cases per million per year.Its mechanisms can be divided into two categories: a decreased production through bone marrow suppression, or an increased destruction through an immune-mediated mechanism. Immune-mediated thrombocytopenia develops generally after 7-14 days of therapy, while non-immune-mediated thrombocytopenia tends to develop more gradually, over a few weeks. Recovery of platelet count occurs several days after disruption of drug administration in immune-mediated thrombocytopenia, while recovery from non immune DIT may take longer.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sepsis having 2 or more of the following criteria:

  1. Septic shock clinically identified by a vasopressor requirement to maintain a mean arterial blood pressure of 65 mm Hg or greater.
  2. Serum lactate level greater than 2 mmol\L.
  3. Positive culture confirming bacterial infection.
* Patients highly susceptible to infection by Gram-positive bacteria such as Nosocomial pneumonia, Community-acquired pneumonia, Complicated skin and soft tissue infections.

Exclusion Criteria:

* Patient or their legal guardian refuses to include their data in the study.
* Known allergy to linezolid.
* Pregnancy and lactation.
* Severe hepatic failure (Child-Pugh C as INR>2.3, Bilirubin>3mg/dl, Albumin<2.8gm/dl).
* Thrombocytopenia (platelet count < 80,000/mm3).
* Disseminated intravascular coagulation (DIC) as Fibrinogen<1g/L, PT more than 6 seconds increase above normal, high D Dimer level.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: After obtaining approval from the research ethical committee of the Anesthesia, Intensive care and Pain management department, Ain Shams University; this study will be conducted in the ICUs of Ain Shams University Hospitals.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
The relationship between kidney function and the development of linezolidinduced thrombocytopenia | Through study completion, an average of 1 year the occurrence of severe thrombocytopenia < 30.000 that will indicate stop receiving medications that implicates in causing thrombocytopenia or transfer of the patient from ICU.

SECONDARY OUTCOMES:
The duration of hospital stay or ICU stay or The incidence of the need for renal replacement therapy (RRT) during hospital stay. | Through study completion, an average of 1 year the occurrence of severe thrombocytopenia < 30.000 that will indicate stop receiving medications that implicates in causing thrombocytopenia or transfer of the patient from ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt